CLINICAL TRIAL: NCT05434533
Title: The Prophylactic Role of Tranexamic Acid in High Risk Pregnant Women Undergoing Elective Cesarean Section in Prevention of Postpartum Hemorrhage
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Hany, MD, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FarahMSc2022
Record Dates: First submitted 2022-06-09; First posted 2022-06-28 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: High Risk Pregnant Women Undergoing Elective Cesarean Section
Keywords: high risk pregnancy; cesarean section.; tranexamic acid
MeSH Terms: interventions — Tranexamic Acid; Adenosine Monophosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- preoperative (Experimental): 1 gm of Tranexamic acid (Kapron, Amoun Pharmaceuticals SAE, Egypt. 5ml Amp, 100mg /1ml) 30 mins before the operation
  Interventions: Drug: Tranexamic acid (Kapron, Amoun Pharmaceuticals SAE, Egypt. 5ml Amp, 100mg /1ml)
- uterine incision (Experimental): 1 gm of Tranexamic acid (Kapron, Amoun Pharmaceuticals SAE, Egypt. 5ml Amp, 100mg /1ml) directly before uterine incision
  Interventions: Drug: Tranexamic acid (Kapron, Amoun Pharmaceuticals SAE, Egypt. 5ml Amp, 100mg /1ml)
- placebo (No Intervention): 1ml of normal saline will be given

INTERVENTIONS:
Drug: Tranexamic acid (Kapron, Amoun Pharmaceuticals SAE, Egypt. 5ml Amp, 100mg /1ml) — IV 1gm
  Arms: preoperative; uterine incision

SUMMARY:
The aim of the study is to assess the prophylactic role of tranexamic acid in reducing blood loss during and after elective cesarean section delivery in high risk patients.

Comparing effect of administration of 1gm of TXA half an hour before elective C-section , effect of administration of 1gm of TXA on the start of uterine incision and placebo effect, Where in all an addition of prophylactic uterotonics is given, in a randomized control, double blind trial of 3 groups.

DETAILED DESCRIPTION:
All patients will undergo the following

I. History : Medical history, Obstetric history, Comorbidities, Allergies. II. Clinically: Vital signs, Abdomino-pelvic examination, per-vaginal examination.

III. Laboratory: Hemoglobin, Hematocrit before & after cesarean section. IV. Routine Ultrasound. V. Cesarean section: done under spinal anathesia.

VI. Calculation of blood loss:

The quantity of blood loss (ml) is calculated from 3 components :

* (weight of used towels during surgery - weight of used towels prior to surgery),plus
* (volume of blood sucked in suction container after placental delivery) ,plus
* (weight of used vaginal pad in the first 2 hours after CS - the pad' s dry weight)
* Each 1 mg increase the weight of either the towels or the vaginal pads is equivalent to 1 ml blood loss (Vitello, Dominic J., et al).

VII. Informed Consent: will be obtained from all participants including the pregnant women who are included in the study .

All patients will receive routine ecbolics ( oxytocin ) after delivery of baby.

ELIGIBILITY:
Inclusion Criteria:

* High risk women undergoing elective C-section

  * Hypertensive patients.
  * Obese patients.
  * Patients on LMWH.
  * Transverse lie
  * DM ( Type 1 & Gestational )
  * Cardiac ( Not on Anticoagulants )
  * Placenta Previa ( Not in PAS )
  * Previous uterine scar ( > previous 2 C- section )

Exclusion Criteria:

* Patients with bleeding tendency.
* HELLP Syndrome.
* Emergency C- section.
* Mechanical prosthetic valve
* Atrial Fibrillation.
* Allery to tranexamic acid
* Placenta Accreta , Increta , percreata.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 156 (Actual)
Dates: Start 2022-07-03 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Reduction of blood loss during C-section. | 1 hour
  ml
Prevention of 1ry postpartum hemorrhage. | 24 hours
  ml

SECONDARY OUTCOMES:
Reduction of hospital stay. | 48 hours
  Number of days
Decrease risk of maternal blood transfusion | 48 hours
  Number of blood products units

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Hany, MD, Principal Investigator — Associate professor
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No